CLINICAL TRIAL: NCT04714645
Title: Effectiveness of Virtual Reality Training on Unilateral Spatial Neglect After Stroke - a Randomized Controlled Trial
Brief Title: Effectiveness of Virtual Reality Training on Unilateral Spatial Neglect After Stroke
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Vrije Universiteit Brussel (Other)
Responsible Party: Principal Investigator, Emma De Keersmaecker, Principal Investigator, Vrije Universiteit Brussel
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VR study - neglect
Record Dates: First submitted 2021-01-11; First posted 2021-01-19 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2022-05

CONDITIONS: Stroke; Neglect
Keywords: virtual reality; neglect; stroke; intervention
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: There will be an external assessor, who will be blinded during the clinical assessments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): VR+ training
  Interventions: Device: VR neglect training
- Control group (Sham Comparator): VR- training
  Interventions: Device: VR control training

INTERVENTIONS:
Device: VR neglect training — Patients will undergo 1 session a day for 30 minutes for 5 consecutive days. The training consists of 5 different VR tasks specifically designed for neglect training.
  Arms: Intervention group
Device: VR control training — Patients will undergo 1 session a day for 30 minutes for 5 consecutive days. This is a placebo training, where patients will also wear the HMD. Patients will be immersed in a virtual environment without a specific task.
  Arms: Control group

SUMMARY:
The aim of this study is to examine the effect of an additional VR training program on unilateral spatial neglect (USN) after stroke. Principally, clinical assessment of the presence of unilateral spatial neglect and additionally the severity of USN will be measured using the Behavioral Inattention test (BIT), using only the BIT Conventional subtest (BITC). Secondarily, the VR outcomes will be included as well.

Finally, we want to determine if the effects last over a short period of time. It is important to know whether the potential effects of the VR-training remain without continuing the intervention. Therefore, we will perform a follow-up assessment after 1 week.

DETAILED DESCRIPTION:
STUDY DESIGN

The design of this study is a 1-week, assessor-blinded randomized controlled trial with a 1-week follow up.

MATERIALS

The HMD VR system 'Oculus Rift' (Oculus, LLS, US) is a low-cost HMD that fully integrates the user into the virtual environment by blocking out perception of the real-world. It includes a headset, two oculus touch controllers and two sensors. To power the Oculus Rift, a compatible laptop will be used. The "Oculus Rift" will assure a fully immersive virtual environment.

PROCEDURE

Pre-treatment assessment: First, eligible patients will be screened and assessed. For screening and assessment, patients will undergo 2 tests: a VR test and a conventional test. The patient will be seated in a (wheel)chair while performing the assessment tests, with one of the researchers present for safety. All patients will immediately complete the tests, without a try-out session. Instructions will be given in a consistent way and during the tests no feedback will be given.

For the VR-test, the HMD will be used. The VR test consists of 5 different tasks:

1. penguin search (1min)
2. smartphone search (1min)
3. apple examination (12 apples)
4. penguin extinction (10 times)
5. grabbing cubes (6 cubes)

For the conventional test, patients will need to perform the Behavioral Inattention test - conventional subtest (BITC), which consists of 6 different tasks:

1. line crossing
2. letter cancellation
3. star cancellation
4. figure and shape copying
5. line bisection
6. representational drawing

Once the assessment is completed, all patients will receive a standard care program provided by the rehabilitation hospital.

Intervention group:

Additionally, the intervention group will receive a VR training for 30 min consisting of various specific developed tasks for unilateral neglect training for a period of five consecutive days (one session a day). The VR training consists of the same 5 tasks used for the assessment. On the last day of the intervention and one week after, patients will be assessed again by completing the BITC test and the VR tasks.

Task 1: Penguin search: the patient has to search a penguin, which is randomly placed in the virtual environment. The patient has to aim for the penguin with this crosshair for a certain amount of time (until the loading bar is filled) in order to receive a point. The penguin is teleported to a new position afterwards. The subject has 2 minutes to gain as many points as possible. When the patient is not able to locate the penguin, arrows will indicate the direction of the penguin.

Task 2: Smartphone search: The Smartphone Search task is similar to the Penguin Search task. This time it takes place in a kitchen and the subject has to search for a smartphone on the kitchen counter. This kitchen counter is located in front of the subject. As in task 1, a crosshair is placed in the center of the camera canvas and the player receives points by aiming at the target. Like before, the subject has 2 minutes to gain as many points as possible. Like in the previous task, some arrows show up after ten seconds to help the subjects when they are not able to find the smartphone.

Task 3: Apple examination: In the Apple Examination task, the patient has to distinguish normal apples from distractors. The subject is placed in a grass landscape with 8 normal apples and 12 distractors. As in the previous tasks, a crosshair is attached to the canvas of the camera. The subject has to aim for the normal apples and press button A or X of the oculus controllers to get a point. The task ends when all normal apples are found.

Task 4: Penguin extinction: This task takes place in the same mountain environment as the Penguin Search task. In contrast with the other tasks, the subject doesn't have to search in the virtual environment, since everything takes place in the subject's field of view. There are three scenario's: either there is one penguin present on the right side, either there is one present on the left, or two penguins are present, one on each side. The subject has to say which scenario was presented by moving the thumbstick of the right or left oculus controller accordingly to the right (correct answer for scenario 1), to the left (correct answer for scenario 2) or upwards (correct answer for scenario 3). A point is gained for every correct answer. The task is completed when the subject has reached a score of thirty.

Task 5: Grabbing cubes: The last task is called Grabbing Cubes. Ten cubes are randomly placed on a table which is located in front of the player. The subjects have to grab the cubes and remove them from the table by dropping them on the ground. Grabbing an object is done by pressing the hand trigger of the left or right oculus controller. In order to complete the task, they have to remove all the cubes from the table.

Control group:

The control group will receive a placebo VR intervention. Patients in the control group will also use the HMD but they will look at another virtual environment with no specific tasks. The virtual environment represents a park outside where other avatars (hikers, joggers) are passing by. Patients will be looking at the environment for the same time as the VR training of the intervention group, i.e. 1 session a day for 5 days. On the last day of the intervention and one week after, patients will be assessed again by completing the BITC test and the VR tasks.

RANDOMIZATION

Participants will be randomly allocated to either the intervention group or the control group (1:1 ratio). Patients will be assigned to a group by block randomization.

STUDY ANALYSIS

Since heterogeneity between groups will be present at baseline, an ANCOVA analysis will be conducted to correct this matter. If significant changes are found at postintervention and follow-up, post-hoc analyses for multiple comparisons will be performed using the Bonferroni correction.

ELIGIBILITY:
Inclusion Criteria:

* a right-hemisphere hemorrhagic or ischemic stroke, confirmed by CT or MRI
* only subacute (>2 weeks) and chronic (>6 months) unilateral spatial neglect patients
* scoring below the cut-off value of 129 points on the standard BITC test
* being 18 years or older at the time of lesion

Exclusion Criteria:

* patients with dementia (Mini Mental State Examination (MMSE) < 24) or aphasia (Mississippi Aphasia Screening Test (MAST) < 45)
* patients whose visual or hearing impairment does not allow possibility of interaction with the VR system
* patients with depression (Patient Health Questionnaire (PHQ-9) >= 10)
* patients unable to sit for at least 30 minutes in a wheelchair or chair
* patients with sensorimotor alterations that can interfere with the performance with the VR system

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-02-15 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
BITC test | through study completion, i.e. 12 days
  The BITC test will be taken before, immediately after and 1-week after the intervention.

SECONDARY OUTCOMES:
VR specific outcome: head rotations | through study completion, i.e. 12 days
  The head rotations (left/right) will be recorded continuously during the VR tasks. The head rotations made during the VR tasks before, immediately after and 1-week after the intervention will be compared
VR specific outcome: time | through study completion, i.e. 12 days
  The time needed to complete the different VR tasks will be recorded. The time needed to complete the VR tasks before, immediately after and 1-week after the intervention will be compared.
VR specific outcome: number of errors | through study completion, i.e. 12 days
  The number of errors made by the patient during the different VR tasks will be recorded. The number of errors made during the VR tasks before, immediately after and 1-week after the intervention will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Eva Swinnen, Prof. Ph.D, Principal Investigator — Vrije Universiteit Brussel
Locations (1):
- Vrije Universiteit Brussel, Brussels, Belgium